CLINICAL TRIAL: NCT00156351
Title: Evaluation of the National Black Women's Health Project Walking for Wellness Program
Brief Title: Walking For Wellness Program Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Shiriki K. Kumanyika, PhD, MPH, RD, University of Pennsylvania
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 707525
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2008-03-28 (Estimated); Status verified 2008-03

CONDITIONS: Physical Inactivity; Obesity
Keywords: African Americans; Women; Internet; Telephone Counseling
MeSH Terms: conditions — Sedentary Behavior; Obesity

INTERVENTIONS:
Behavioral: Physical activity promotion

SUMMARY:
The overall purpose of this project is to conduct an innovative, culturally-tailored demonstration project designed to facilitate the adoption and maintenance of regular, moderate physical activity (i.e., brisk walking) in a sample of sedentary African American women. In addition, we will test the impact of varying types of counseling and social support on the adoption and maintenance of regular physical activity and help women improve their weight control. The core behavioral change program will be based on a comprehensive wellness oriented website offered by the National Black Women's Health Project (NBWHP). Comparisons will be made between the effects of the web-based program with only minimal face to face contacts, primarily for enrollment, data collection, and participant retention, the web-based program with the addition of telephone counseling and support, and the web-based program with face to face group counseling and support.

Hypotheses. Hypothesis 1. Participation in the intervention will result in increased physical activity levels, regardless of the level of social support.

Hypothesis 2. The intervention arm involving the lowest level of social support will be marginally effective for increasing physical activity levels, and additional social support will result in significantly improved physical activity levels when compared with the lowest level of social support.

The specific intervention questions are:

1. How well do the interventions address the program objectives ((quality of implementation), to be determined through protocol review for operationalization of theoretical constructs)?
2. Was the program implemented as planned ((fidelity to protocol and dose of intervention), to be determined from implementation process variables, including characteristics of women recruited, fidelity to protocols for contact with participants, and quality of counseling given, where applicable)?
3. Did the program (separately for each format tested) have a significant effect on potential mediators of behavior change (influence on presumed intermediate outcomes)? For the purpose of this proposal, a mediator is defined as any barrier to or facilitator of physical activity participation (e.g., time, self efficacy, social support, access, perceived norms) as implied in the 12 behavioral objectives that have been specified.
4. What is the optimum type of counseling and support to enhance the on-line activities in order to produce significant behavior change (importance of various program components)?
5. Did the program (separately for each format tested) have a significant effect on the primary study outcomes (influence on primary behavioral outcome, e.g., physical activity by self-report of activity levels or pedometer counts)?
6. Do changes in mediators explain changes in the primary outcomes (multivariate models to understand if presumed process of behavioral change was observed in practice)?
7. Does the internet only program appear to result in increased physical activity participation when compared to extant data on trends among Black women in the U.S. population (what is accomplished with very minimal intervention and how does it compare with a more extensive program)?

ELIGIBILITY:
Inclusion Criteria:

* African American Women
* 18 years of age and older
* Have a working telephone
* Have reliable internet service

Exclusion Criteria:

* Men
* Physical limitations and/or disabilities that would preclude a walking program
* Report currently meeting the minimum physical activity guidelines, as they relate to health and/or weight loss

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186
Dates: Start 2003-01; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Physical activity level

CONTACTS AND LOCATIONS:
Overall Officials: Shiriki K Kumanyika, PhD, MPH, RD, Principal Investigator — University of Pennsylvania
Locations (1):
- 3401 Market Street, Suite 202, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Related Info — http://www.blackwomenshealthimperative.org